CLINICAL TRIAL: NCT05446090
Title: Asthma: Phenotyping Exacerbations 3
Acronym: APEX3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 304615-21066
Record Dates: First submitted 2022-05-26; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Asthma Attack
MeSH Terms: interventions — Fractional Exhaled Nitric Oxide Testing; Nasal Absorption; Health Records, Personal; Demography; Sino-Nasal Outcome Test; 4-amino-4'-hydroxylaminodiphenylsulfone; Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and sputum samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Asthma Attack patients.: Patients admitted with Asthma Attacks.
  Interventions: Diagnostic Test: Spirometry including peak flow; Diagnostic Test: Fractional Exhaled Nitric Oxide (FeNO); Diagnostic Test: Forced Oscillation Technique (FOT); Procedure: Sputum Induction; Diagnostic Test: Bloods; Diagnostic Test: Nasal lavage; Diagnostic Test: Throat swab; Diagnostic Test: Nasal Brush.; Diagnostic Test: Nasal absorption; Other: Medical History, Demographic, and Concomitant Medications; Other: Sino-nasal Outcome Test; Other: Gastroesophageal Reflux Disease Questionnaire; Other: Pittsburgh Vocal Cord Dysfunction Index; Other: Nijmegen Questionnaire.; Other: Hospital Anxiety and Depression Scale; Other: Compliance and adherence; Other: Acute Asthma Quality of Life Questionnaire

INTERVENTIONS:
Diagnostic Test: Spirometry including peak flow — Spirometry including peak flow to assess the degree of airway obstruction. Spirometry will be conducted according to a study SOP. The Global Lung Function (GLI) 2012 equations will be used. Reversibility testing will not be routinely performed. Thus, asthma medications will not normally be withheld for study visits and patients should take their inhalers as usual. The same type of device will be used at each visit.
Diagnostic Test: Fractional Exhaled Nitric Oxide (FeNO) — Fractional Exhaled Nitric Oxide (FeNO) to assess the degree of airway inflammation. FeNO will be measured using a standard device (NIOXX Vero®) in accordance with the manufacturer's guidelines. The same type of device will be used at each visit. FeNO should be performed prior to any other respiratory assessment if possible.
Diagnostic Test: Forced Oscillation Technique (FOT) — FOT is a non-invasive method that evaluates resistance and reactance in the respiratory system during tidal breathing. It should be performed after FeNO, but prior to Spirometry and will be conducted according to a study SOP.
Procedure: Sputum Induction — Sputum Induction for the assessment of airway inflammation and microbiology. Sputum induction will be performed according to an SOP, which includes measures to protect the safety of participants. These consist of pre-treatment with Salbutamol, a short acting bronchodilator, stipulated levels of lung function in order to perform the test and stopping criteria. If the participant is unable to undergo the procedure, due to safety reasons, they will be asked to produce a spontaneous sputum sample. Sputum samples will be collected for a differential cell count, bacterial culture and sensitivity and storage for future research. Procedures for sampling and processing will be detailed in a study SOP.
Diagnostic Test: Bloods — Blood will be collected for laboratory analysis, including Vitamin D, Haematology, WCC differential, C-Reactive protein.
Diagnostic Test: Nasal lavage — Nasal lavage samples will be taken at the baseline (attack) visit. Samples will be obtained by injecting 5ml of sterile normal saline into the participant's nostrils via a nasal adaptor and then immediately aspirated. These will be placed in a sterile container and transported to the laboratory for viral identification. This procedure will be detailed in a study SOP.
Diagnostic Test: Throat swab — A throat swab will be taken at the baseline (attack) visit for viral identification.
Diagnostic Test: Nasal Brush. — Nasal brushings samples may be taken at baseline (attack) and at second visits for RNA and DNA extraction. This will be optional and specific consent from participants will be sought. Procedures for sampling and processing will be detailed in a study SOP.
Diagnostic Test: Nasal absorption — Nasal absorption will be used to collect mucosal lining fluid from the respiratory tract for cytokines profiling at baseline (attack) and at second visits.
Other: Medical History, Demographic, and Concomitant Medications — Medical history will include clinically significant diseases and prior surgeries and smoking history. A specific respiratory history will also be recorded. Demographic data will include age, sex and self- reported race/ethnicity. Medication use will also be collected.
Other: Sino-nasal Outcome Test — The incidence of upper airway symptoms will be assessed using Sino-nasal Outcome Test (SNOT).
Other: Gastroesophageal Reflux Disease Questionnaire — The incidence of Gastroesophageal Reflux Disease will be assessed using GERDQ questionnaire.
Other: Pittsburgh Vocal Cord Dysfunction Index — The incidence of vocal cord dysfunction will be assessed using Pittsburgh Vocal Cord Dysfunction (VCD) Index
Other: Nijmegen Questionnaire. — The incidence of dysfunctional breathing will be assessed using Nijmegen dysfunctional questionnaire.
Other: Hospital Anxiety and Depression Scale — The incidence of anxiety and depression will be assessed using Hospital Anxiety and Depression Scale (HADS).
Other: Compliance and adherence — In order to assess adherence as a factor in exacerbations, a participant's beliefs and attitudes towards medicines will be explored using the Medicines Adherence Report Scale (MARS) questionnaire. Non-intentional non-compliance with usual treatment will be assessed by checking inhaler technique; poor inhaler technique will be reported to the participant's clinical team. Also, GP records will be reviewed for information on medications prescribed in the last 12 months.
Other: Acute Asthma Quality of Life Questionnaire — The impact of acute asthma on quality of life will be assessed using Acute Asthma Quality of Life Questionnaire at baseline and follow up.

SUMMARY:
Exacerbations of asthma (asthma attacks) are very common in the UK. They are frightening for patients, expensive for the health service, and occasionally lead to avoidable deaths.

Despite the obvious importance of asthma attacks, they remain poorly understood. Although some of the triggers for attacks are known, the resultant characteristics of attacks are not. Recent research has shown different inflammation profiles associated with asthma attacks; however, this is not well understood, and all asthma attacks are treated the same. Increased knowledge about the nature of asthma attacks may better define these attacks and help develop more targeted treatment options.

This study aims to describe the characteristics of patients admitted with asthma attacks. The recovery and response to standard treatment for asthma attacks following discharge from the hospital will also be described.

This is achieved by studying the characteristics of asthma attacks in patients hospitalized with acute asthma. Participants will be asked to attend two follow-up visits during which their response to treatment will be described.

The study is planned to last for 2.5 years, with a recruitment period of 18 months, and will include 100 participants with acute asthma.

DETAILED DESCRIPTION:
Asthma is a common condition affecting 9.8 million people in the United Kingdom1. Asthma attacks cause nearly 1500 deaths per year in the UK2 and account for over 90,000 hospital admissions and 1800 intensive care admissions costing at least 1 billion pounds a year3.

Non-asthma conditions such as Vocal Cord Dysfunction4 and Dysfunctional Breathing Pattern5 can mimic severe asthma and lead to hospital admission and inappropriate asthma treatment with potentially harmful high dose corticosteroids. However, the proportion of patients admitted with these asthma mimics is unclear.

The use of biomarkers to guide treatment in stable asthma is now commonplace, but this prospect has not been fully explored in acute asthma attacks. Determining the type of inflammation underlying an attack can, however be tricky because many patients receive oral corticosteroid prior to, or soon after admission, which promptly and markedly affects the most accessible type 2 asthma (T2) biomarkers7, the blood eosinophil count. Measurement of another T2 biomarker, fractional exhaled nitric oxide (FENO), during an attack may prove a useful measure of ongoing T2 airway inflammation, but this strategy requires assessment.

Airway obstruction in asthma attacks is assessed and confirmed by measuring peak expiratory flow and/or forced expiratory volumes. These measures are effort-dependent and can, therefore, be unreliable and misleading if improperly performed. We aim to evaluate the potential feasibility and utility of alternative diagnostic methods of assessing airway obstruction and measuring T2 biomarkers to see if these allow the distinction between actual asthma attacks and asthma attack mimics and also if they can distinguish different types of asthma attacks.

The pattern of recovery following asthma attacks is also not fully understood. Studies have reported varying recovery times8 and inconsistencies in the response of airway obstruction9 and T2 biomarkers10 to corticosteroid treatment in acute asthma.

The investigators hypothesise that a significant proportion of patients admitted to hospital with suspected asthma attacks have an alternate cause for their clinical presentation. To further explore this, The investigators propose an observational study to describe and investigate the characteristics of patients admitted with suspected severe asthma. The investigators will assess the utility of point of care, non-invasive biomarker measurements in identifying pulmonary and extrapulmonary traits in patients hospitalised due to presumed asthma attack. A variety of study assessments will be performed at the baseline visit (exacerbation visit), and two follow up visits following hospital discharge. Results of study assessments obtained during each study visit will be compared and analysed. This is the first study to prospectively investigate acute asthma both during and following exacerbation episodes. This will allow a comprehensive understanding and description of pulmonary and extrapulmonary traits as well as the pattern of recovery following asthma attacks.

ELIGIBILITY:
Inclusion Criteria:

* The ability to give fully informed consent
* Male or female aged ≥ 18 years of age.
* Admission with a suspected acute asthma attack.
* Able (in the investigator's opinion) and willing to comply with clinical investigation requirements.

Exclusion Criteria:

* Other clinically significant respiratory diseases including predominant Chronic Obstructive Pulmonary Disease (COPD) and bronchiectasis.
* Any other clinically significant medical disease or uncontrolled concomitant disease that is likely, in the investigator's opinion, to impact the ability to participate in the study or the study results.
* Pregnant women, lactating women or women who are planning to become pregnant.
* Investigator determined apparent other cause for admission.
* Acute COVID infection.
* Non-English-speaking participants who are unable to comprehend the reasons for the study due to limitations in understanding the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with suspected asthma attacks.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of cytokine levels in nasal lining fluid at attack and recovery visits | 14 days
  Nasal absorption will be used to collect mucosal lining fluid from the respiratory tract for cytokines profiling at baseline (attack) and at second visits.
The measurement of vitamin D levels in the blood on admission to the hospital | baseline
  vitamin D levels in the blood on admission to the hospital
Assessment of evidence of infection: sputum for bacterial culture and sensitivity (MC&S). | 14 days
  Assessment of evidence of infection: sputum for bacterial culture and sensitivity (MC&S).
Assessment of evidence of infection: CRP. | 14 days
  Assessment of evidence of infection: CRP.
Assessment of evidence of infection: Throat swab/nasal lavage for viral PCR. | baseline
  Assessment of evidence of infection: Throat swab/nasal lavage for viral PCR.
A specific asthma history (polypharmacy, previous asthma attacks, triggers, Personalised Asthma Action Plan) for the assessment of risk factor for attack. | baseline
  Assessment of risk factor for attack
Assessment of adherence to medications (MARS, prescription records, inhaler technique) for the assessment of behavioural attack traits. | baseline
  Assessment of behavioural attack traits.
Assessment of airway obstruction at attack and recovery visits using peak expiratory flow rate (PEFR). | 14 days
  Assessment of airway obstruction
Assessment of airway obstruction at attack and recovery visits using spirometry. | 14 days
  Assessment of airway obstruction
Assessment of airway obstruction at attack and recovery visits using Forced Oscillation Technique (FOT). | 14 days
  Assessment of airway obstruction
Assessment of airway obstruction at attack using physician recorded expiratory wheeze | baseline
  Assessment of airway obstruction
Assessment of airway inflammation at attack and recovery visits using Fractional Exhaled Nitric Oxide (FeNO). | 14 days
  Assessment of airway inflammation
Assessment of airway inflammation at attack and recovery visits using sputum inflammatory cell count. | 14 days
  Assessment of airway inflammation
Assessment of airway inflammation at attack and recovery visits using blood eosinophil count. | 14 days
  Assessment of airway inflammation
Assessment of symptom burden at attack and recovery visits using the Acute AQLQ questionnaire | 28 days
  Assessment of symptom burden
Assessment of Body Mass Index BMI. | baseline
  Assessment of Body Mass Index BMI.
Assessment of the incidence of upper airway symptoms. | baseline
  The incidence of upper airway symptoms will be assessed using the Sino-nasal Outcome Test (SNOT).
The assessment of the incidence of Gastroesophageal Reflux Disease. | baseline
  The assessment of the incidence of Gastroesophageal Reflux Disease using the GERDQ questionnaire.
The assessment of the incidence of vocal cord dysfunction | baseline
  The assessment of the incidence of vocal cord dysfunction using the Pittsburgh Vocal Cord Dysfunction (VCD) Index.
The assessment of the incidence of dysfunctional breathing | baseline
  The assessment of the incidence of dysfunctional breathing using the Nijmegen dysfunctional questionnaire.
The assessment of the incidence of anxiety and depression | baseline
  The assessment of the incidence of anxiety and depression using the Hospital Anxiety and Depression Scale (HADS).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Martin, Principal Investigator — The University of Nottingham
Locations (1):
- Nottingham University Hospital, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
No plans yet.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT05446090/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT05446090/ICF_001.pdf